CLINICAL TRIAL: NCT02355704
Title: Anti-inflammatory Effect of Atorvastatin on Graft Donor Kidney Transplantation in Vivo
Brief Title: Anti-inflammatory Effect of Atorvastatin on Graft Donor Kidney
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, CLOTILDE FUENTES OROZCO, PhD, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-1301-78
Record Dates: First submitted 2015-01-22; First posted 2015-02-04 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-01

CONDITIONS: Renal Insufficiency
Keywords: Kidney Transplantation; Atorvastatin; C-Reactive Protein; Biopsy; Interleukin
MeSH Terms: conditions — Renal Insufficiency | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Active Comparator): 22 patients received oral atorvastatin 40 mg 1 time for day for 4 weeks
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): 22 patients received oral placebo 40 mg 1 time for day for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Patients were assigned to two groups, one of them received oral atorvastatin (study group) and the other, homologated placebo (control group) for 4 weeks before a kidney transplantation. Previous surgical procedure controls were performed
  Other Names: Lipitor
  Arms: Atorvastatin
Drug: Placebo — Patients were assigned to two groups, one of them received oral atorvastatin (study group) and the other, homologated placebo (control group) for 4 weeks before a kidney transplantation. Previous surgical procedure were performed
  Other Names: Homologated Placebo
  Arms: Placebo

SUMMARY:
Renal Insufficiency is a priority disease in health system, which may require renal replacement therapy based on renal transplantation, which is considered as therapy of choice. During the procedure of renal transplantation, the graft could be damaged by ischemia-reperfusion which generates complications in its function.

Recently the anti-inflammatory and immunomodulatory effects of statins have been emphasized, which could be beneficial in renal transplantation.

DETAILED DESCRIPTION:
Objective: Evaluate anti-inflammatory effect of atorvastatin on renal graft in living donor transplantation.

Material and methods: Controlled, double-blind clinical trial with posterior following for 12 months. Composed by 48 patients, randomized manner, realized at the Transplant Department of Western Medical Center, Mexican Institute of Social Security. Universe was patients accepted as kidney donors. Patients were randomized in two groups (study or control) the intervention was implemented 4 weeks before kidney transplant. Previous surgical procedure, in a blood sample, C-Reactive Protein (C-RP) and laboratory control were measured. During surgical procedure, a biopsy was obtained to measure IL-6 and tumoral necrosis factor alpha by immunohistochemistry. 24 hours after surgical procedure, 3 and 12 months of following, kidney function, complications and graft survival were registered. During surgical procedure, 3 months and 12 months of following, biopsies were obtain to performed histopathological analysis of scale of Banff

The statistical analysis was performed according to the nature of variables, for continuous data using measures of central tendency and dispersion and for the qualitative data with frequencies and percentages.

ELIGIBILITY:
Inclusion Criteria:

* Accepted as kidney donor
* Voluntary participation
* Informed consent accepted
* 85% fulfillment of atorvastatin treatment

Exclusion Criteria:

* Hypersensibility to Atorvastatin
* Smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-01; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
C-Reactive Protein evolution in donors | Basal and 4 weeks later
  C-Reactive Protein was measured when patients (donors) were accepted in the study and 4 weeks later. The last blood sample was taken the day of surgical procedure.
Kidney graft rejection using scale of BANFF | Basal, 3 months and 12 months
  During surgical procedure and before organ transplantation, basal biopsy was obtain. In the following at 3 and 12 months after kidney transplantation, were performed the other two biopsy. Alterations between groups were registered.

SECONDARY OUTCOMES:
Kidney function evolution after transplant | 24 hours, 3 months and 12 months
  In blood samples, after kidney transplantation, creatinine and urea were measured. Differences in evolution and alteration between the 2 groups were registered
Interleukin and tumor necrosis factor alpha. | Basal
  During surgical procedure and before organ transplantation, the biopsy was obtain to measure interleukin 6 and tumor necrosis factor alpha, observing alteration between groups.
Complications | 24 hours, 3 months and 12 months
  During surgical procedure, any kind of complication was registered, the same right after surgery and in the following.

CONTACTS AND LOCATIONS:
Overall Officials: Clotilde Fuentes-Orozco, PhD, Study Director — Instituto Mexicano del Seguro Social
Locations (1):
- Western Medical Center, Mexican Institute of Social Security, Guadalajara, Jalisco, Mexico